CLINICAL TRIAL: NCT02687477
Title: Pulmonary Artery Denervation to Treat Severe Obstructive Sleep Apnea: a Single-center, Prospective, First-in-man Study（PADN-OSA）
Brief Title: PADN to Treat Severe Obstructive Sleep Apnea
Acronym: PADN-OSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients meeting the criteria for admission
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFH20160106
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham procedure (Sham Comparator): Patients in the sham group will take sham procedure like PADN.
  Interventions: Procedure: Sham procedure
- Pulmonary Arterial Denervation (Experimental): Contrast pulmonary artery （PA) angiography was performed to localize the pulmonary artery bifurcation level and calculate the PA diameter.Once the anatomy was deemed acceptable, the radiofrequency ablation catheter was introduced into the distal bifurcation area of the main PA.This was then maneuvered within the PA to allow energy delivery to ensure that the electrodes were tightly in contact with the endovascular surface. About two to three ablations at 1-15 W for 240 seconds each point were performed in the distal bifurcation area of the main PA.
  Interventions: Procedure: Pulmonary Arterial Denervation

INTERVENTIONS:
Procedure: Pulmonary Arterial Denervation — Contrast pulmonary artery （PA) angiography was performed to localize the pulmonary artery bifurcation level and calculate the PA diameter.Once the anatomy was deemed acceptable, the radiofrequency ablation catheter was introduced into the distal bifurcation area of the main PA.This was then maneuvered within the PA to allow energy delivery to ensure that the electrodes were tightly in contact with the endovascular surface. About two to three ablations at 1-15 W for 240 seconds each point were performed in the distal bifurcation area of the main PA.
  Arms: Pulmonary Arterial Denervation
Procedure: Sham procedure — patient in the sham group will receive sham procedure
  Arms: Sham procedure

SUMMARY:
This project is focused on the treatment of severe obstructive sleep apnea with pulmonary artery denervation (PADN). Although it has now been proved that continuous positive airway pressure (CPAP) is the primary treatment for obstructive sleep apnea, on the other hand, there is evidence that 25 to 50% of patients can not tolerate CPAP.

The investigators previously reported the safety and efficacy of pulmonary artery denervation (PADN) for treatment of pulmonary hypertension. Excessive sympathetic activation play an important role in the occurrence and development of OSA and cause cardiovascular events. It is worth evaluating the feasibility and tolerance of introducing PADN at the severe stage of obstructive sleep apnea. Therefore, the purpose of our study is to evaluate the safety and feasibility of PADN in the treatment of severe OSA.

ELIGIBILITY:
Inclusion Criteria:

* Apnea hypopnea index more than 30, not tolerated or refused continuous positive airway pressure;

Exclusion Criteria:

* Acute coronary syndrome;
* Pregnant;
* Expected life less than 12 months;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02; Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
the change from baseline to month 6 in apnea-hypopnea index | Baseline and 6 months

SECONDARY OUTCOMES:
the absolute change in Epworth Sleepiness Scale from baseline to follow-up | Baseline and 6 months

OTHER OUTCOMES:
the change in obstruction of the upper airway by MRI scan | Baseline and 6 months
the change in interleukin-6 (IL-6) at 6-month follow-up | Baseline and 6 months
the change in C-reactive protein at 6-month follow-up | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China